CLINICAL TRIAL: NCT04174040
Title: The Effect of Gross' Process Model of Emotion Regulation Integrated in Musical Rhythm Interventions on Student Nurses' Anger Expressions and States
Brief Title: Process Model of Emotion Regulation Integrated Musical Rhythm Interventions' Effects on Student Nurses' Anger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gizem Beycan Ekitli, PhD., Research Assistant, Ege University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: EgeTrial
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Anger
Keywords: music; Cognitive Behavioral Therapy; randomized controlled trial; rhythm

STUDY DESIGN:
Intervention Model Description: One experimental and three control groups involved study model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control 1 (No Intervention): Applied any intervention.
- Control 2 (Active Comparator): Gross's Process of Emotion Regulation Model interventions applied.
  Interventions: Behavioral: Gross's Process of Emotion Regulation Model Interventions
- Control 3 (Active Comparator): Musical rhythm interventions applied.
  Interventions: Behavioral: Musical Rhythm Interventions
- Experimental (Experimental): Musical rhythm integrated Gross's Process of Emotion Regulation Model interventions applied.
  Interventions: Behavioral: Gross's Process of Emotion Regulation Model Interventions; Behavioral: Musical Rhythm Interventions; Behavioral: Musical Rhythm Integrated Gross's Emotion Regulation Process Interventions

INTERVENTIONS:
Behavioral: Gross's Process of Emotion Regulation Model Interventions — Interventions were based on Gross's Process Model which include the basis concepts of cognitive-behavioral therapy and carried on with five semi-structured sessions. Cognitive-behavioral theories accept the existence of a thought process (attention-perception-interpretation) that appears in the mind about the event just before the anger emerges. Therefore, anger studies with cognitive-behavioral approach generally proceed with the steps of gaining awareness about this concealed thought, identifying behavioral response and avoidance attitudes and thus regulating emotion. It consists of five 90-minute group sessions structured in this context. While being an accredited cognitive behavioral therapist, investigator have qualified to manage these approach.
  The effectiveness of these semi-structured sessions were evaluated by using:
  1. Pretest application of STAXI
  2. Taking feedback after each intervention session
  3. Posttest application of STAXI
  4. Follow-up test application of STAXI
  Arms: Control 2; Experimental
Behavioral: Musical Rhythm Interventions — This musical group rhythm intervention was continued with 90 minute long five sessions. The students participated in the practice together with a music expert and lead researcher. The lead researcher took on the role of observer in these sessions. Each session was continued with warming, improvisation and targeted semi-structured rhythm practices aiming anger regulation. The effectiveness of these semi-structured sessions were evaluated by using:
  1. Pretest application of STAXI
  2. Taking feedback after each intervention session
  3. Posttest application of STAXI
  4. Follow-up test application of STAXI
  Arms: Control 3; Experimental
Behavioral: Musical Rhythm Integrated Gross's Emotion Regulation Process Interventions — The students participated in the practice together with a music expert and lead researcher. The lead researcher ensured the integration of rhythm applications into the Process Model through cognitive-behavioral semi-structured interventions. Five semi-structured 90-minute group sessions were performed. The effectiveness of the experiment was evaluated by using:
  1. Pretest application of STAXI
  2. Taking feedback after each intervention session
  3. Posttest application of STAXI
  4. Follow-up test application of STAXI
  Arms: Experimental

SUMMARY:
Aim: The study aims to determine the effect of the anger management program to be implemented by integrating the rhythm component of music with the Gross Process Model of Emotion Regulation on the anger expression and anger types of nursing students determined to be under risk through screenings.

Materials and Methods: This single-blind factorial designed randomized experimental research was conducted with three control groups. The study group consisted of third-grade students (N=67) who were determined to have scores above average from The State-Trait Anger Expression Inventory (STAXI). The study data were collected with pre-post tests and follow-up measurements using STAXI. The experimental interventions were completed in five sessions after pilot study with a specialist. The data were analyzed using one-way and two-way variance analyses (4x3 Factorial ANOVA). Effect size was measured with ε^2.

DETAILED DESCRIPTION:
Introduction: Nursing students' anger regulation functionally has increasingly gained importance. It is known that cognitive behavioral approaches and music can be used as effective tools for young adults. It is important that the rhythm component of music be integrated with the Gross Model of Emotion Regulation, which analyzes the emotional regulation processes on a cognitive-behavioral basis, and new interventional tools be developed, which can be regularly and easily accessed in psychiatric nursing. The study results will shed light on future studies in terms of using the Gross Model, integrated in musical rhythm studies, to manage functional anger in student nurses.

Aim: The study aims to determine the effect of the anger management program to be implemented by integrating the rhythm component of music with the Gross Model of Emotion Regulation on the anger expression and anger types of nursing students determined to be under risk through screenings.

Materials and Methods: This single-blind factorial designed randomized experimental research was conducted with three control groups. The study group consisted of third-grade students (N=67) who were enrolled in Ege University Faculty of Nursing and determined to have scores above average from The State-Trait Anger Expression Inventory (STAXI). The study data were collected from 38 students who met the inclusion criteria. They were collected with pre-post tests and follow-up measurements using STAXI and introductory information form developed in light of the literature. The Gross Model of Emotion Regulation intervention program, integrated with musical rhythms, was completed in five sessions after pilot study. The sessions in the musical rhythms were carried out in company with a specialist. The data were analyzed using one-way and two-way variance analyses (4x3 Factorial ANOVA). The statistical significance level was measured with p˂0.05, and effect size was measured with ε^2. Ethical permissions were obtained to conduct the study.

ELIGIBILITY:
Inclusion Criteria:

* To be a third year student in the Faculty of Nursing
* To have a higher score than the average limits calculated according to the State Anger score to be obtained from all students,
* Willingness and volunteering for a musical practice

Exclusion Criteria:

* To benefit from regular psychological counseling in the last three months,
* To have a professional music education,
* To have a physical handicap that will affect musical sense and skill.

Ages: 20 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Anger State and Anger Expressions (first evaluation with posttest) | Through study completion, an average of 4 months
  Anger state and expressions were evaluated with using The State-Trait Anger Expression Inventory. This scale originally organized by Charles D. Spielberger in 1988. The scale, which evaluated trait anger (10 items) and state anger behavior (24 items), was adapted to Turk society by Özer N. in 1992. This tool was used to diagnose anger severity and behavioral reactions of anger in many national studies in child, adolescent and adult groups. Scale's Trait Anger dimension (anger expressions) were separated in three subscales as 'anger out', 'anger in' and 'anger control' which each includes eight items (subscale total score min:8, max:32). State Anger subscale has 10 items and total score range is between 10-40 points.
Anger State and Anger Expressions (second evaluation with follow up) | Through study completion, an average of 7 months
  Anger state and expressions were evaluated with using The State-Trait Anger Expression Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Beycan Ekitli, PhD, Principal Investigator
Locations (1):
- Ege University Faculty of Nursing, Izmir, Turkey (Türkiye)